CLINICAL TRIAL: NCT03467256
Title: A Single-Arm Phase I/II Study Evaluating the Safety and Clinical Efficacy Of the 2-nd Generation CD19 Autologous CAR T Cells on the CliniMACS Prodigy Automated Manufacturing Platform in Treatment of Paediatric And Young Adult Patients With Relapsed/Refractory B-lineage Acute Lymphoblastic Leukemia
Brief Title: CD19 T-CAR for Treatment of Children and Young Adults With r/r B-ALL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCPHOI-2018-01
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; Acute Lymphocytic Leukemia, Pediatric
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Immunotherapy, Adoptive; fludarabine; Cyclophosphamide; tocilizumab; Cytarabine; Etoposide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental): Patients will receive lymphodepleting chemotherapy, one hour prior to infusion of CAR T-cells patients will receive tocilizumab IV 8 mg/kg (max 800 mg) over 1 hour. Patients then receive CD19-CAR T cells IV on day 0.
  Interventions: Biological: Chimeric Antigen Receptor T-Cell Therapy; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Tocilizumab; Drug: Cytarabine; Drug: Etoposide; Drug: Dexamethasone

INTERVENTIONS:
Biological: Chimeric Antigen Receptor T-Cell Therapy — anti-CD19 chimeric antigen receptor - transduced T-cell given IV
Drug: Fludarabine — given IV
Drug: Cyclophosphamide — given IV
Drug: Tocilizumab — given IV
Drug: Cytarabine — given IV
Drug: Etoposide — given IV
Drug: Dexamethasone — given IV

SUMMARY:
The purpose of this study is to evaluate the safety and efficiency of autologous CD19 CAR-T lymphocytes in a cohort of pediatric and young adult patients with relapsed /refractory B-lineage acute lymphoblastic leukemia

DETAILED DESCRIPTION:
The main objectives of the study are:

1. To investigate the safety of auto-CD19 CAR T-cells therapy among children and young adults with refractory/relapsed B-cell ALL on the basis of prospective evaluation of adverse affects frequency and severity according to CTCAE v.4
2. To study the efficacy of auto-CD19 CAR T-cells therapy among children and young adults with refractory/relapsed B-cell ALL on the basis of proportion of patients in haematological and molecular remission at 28 days after infusion.
3. To evaluate long-term efficacy of auto-CD19 CAR T-cells therapy among children and young adults with refractory/relapsed B-cell ALL on the basis of overall and event-free survival at 1 and 3 years after infusion.

The novelty of this study will be cytokine release syndrome prophylaxis by tocilizumab Patients will receive fludarabine 120 mg/m2 (totally) intravenously (IV) over 30 minutes on days -5 to -2 and cyclophosphamide 750 mg/m2 IV over 60 minutes on day -2. One hour prior to infusion of CAR T-cells patients will receive tocilizumab IV 8 mg/kg (max 800 mg) over 1 hour. Patients then receive CD19-CAR T cells IV over 20-30 minutes on day 0.

This is a dose-escalation study of CD19-CAR T cells. Dose escalation consistently:

* Level 1 5х105/kg CD19 CAR-T lymphocytes
* Level 2 1х106/kg CD19 CAR-T lymphocytes
* Level 3 3х106/kg CD19 CAR-T lymphocytes
* Level 0 1х105/kg CD19 CAR-T lymphocytes (in case of dose-limiting toxicity at dose Level 1) In case of severe side affects next dose will be reduced to the previous lower dose.

Based on interim analysis the following dosing approach based on stratification by the initial leukemia burden will be implemented starting November 2019:

• Patients with low disease burden (<15% blast cells in BM) will receive a lymphodepletion chemotherapy of fludarabine IV (total dose 120mg/m2) and cyclophosphamide IV (total dose 750mg/m2) over 5 days.

CD19 CAR-T cells will be infused IV in dose 1x106/kg on day 0.

• Patients will high disease burden (>15% blast cells in BM) will receive a lymphodepletion chemotherapy of fludarabine IV (total dose 120 mg/m2), cyclophosphamide IV (total dose 750 mg/m2), cytarabine IV (total dose 900 mg/m2), etoposide IV (total dose 450 mg/m2), dexamethasone IV (total dose 30 mg/m2) over 5 days.

CD19 CAR-T cells 1st dose will be infused IV on day 0 - 0,1x106/kg, 2nd dose will be infused IV between day 7 and 14 - 0,9x106/kg.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent (for patients > 14 years old). For subjects < 18 years old their legal guardian must give informed consent
* Patients with relapsed or refractory CD19-expressing B cell ALL :

  * Induction failure, no CR after course 2 or MRD>0,1% after 3 courses of high-risk protocol
  * early bone marrow or combined relapse of acute lymphoblastic leukaemia, no CR or MRD>0,1% after 1 course 2-nd line therapy
  * ALL post ≥ 2nd relapse, no CR or MRD>0,1% after 1 course 2-nd line therapy
  * Relapse or MRD >0,1% of ALL after stem cell transplant (> 60 days post alloHSCT)
  * Late bone marrow or combined relapse of acute lymphoblastic leukaemia, no CR or MRD>0,1% after 2nd course of 2-nd line therapy
* There must be no available alternative curative therapies
* CD19 expression must be detected on greater than 30% by flow cytometry
* Patients must have measurable or evaluable disease at the time of enrolment, which may include any evidence of disease including minimal residual disease detected by flow cytometry, cytogenetics, or polymerase chain reaction (PCR) analysis.
* Patient Clinical Performance Status: Karnofsky >50% or Lansky >50%
* Patient Life Expectancy > 8 weeks
* Patients recovered from acute toxic effects of all prior chemotherapy, immuno- or radiotherapy
* Patient absolute lymphocyte N > or =100/mm3
* Patient cardiac function: left ventricular ejection fraction greater than or equal to 40% by MUGA or cardiac MRI, or fractional shortening greater than or equal to 28% by ECHO or left ventricular ejection fraction greater than or equal to 50% by ECHO.
* Patients who agree to long-term follow up for up to 5 years (if received CD19 CAR-T cell infusion)

Exclusion Criteria:

1. <30% expression of CD19 on the leukemic population
2. Active hepatitis B, C or HIV infection
3. Oxygen saturation < or = 90%
4. Bilirubin >3x upper norma limit
5. Creatinine >3x upper norma limit
6. Active acute GVHD overall grade ≥2 (Seattle criteria)
7. Moderate/severe chronic GVHD (NIH consensus) requiring systemic steroids
8. Clinical signs of grade >3 CNS disorders (seizure disorder, paresis, aphasia, cerebrovascular, ischemia/hemorrhage, severe brain injuries, dementia, cerebellar disease, organic brain syndrome, psychosis, coordination or movement disorder)
9. Pregnant or lactating women.
10. Active severe infection

Ages: 3 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-05-14 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3-5 SAE occurring within 30 days of CD19CAR T-cell infusion | 1 month
  incidence of grade 3-5 SAE according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 occurring within 30 days of CD19CAR T-cell infusion
Incidence of grade 3-4 Severe Cytokine Release Syndrome following CD19 CAR T-cell infusion | 1 month
  incidence of grade 3-4 Severe Cytokine Release Syndrome
Incidence of grade 3-5 neurotoxicity occurring within 30 days of CD19 CAR T-cell infusion | 1 month
  incidence of grade 3-5 neurotoxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 occurring within 30 days of CD19 CAR T-cell infusion
Proportion of patients in MRD-negative remission | 1 month
  Proportion of patients in MRD-negative remission among all enrolled patients
Proportion of patients in hematologic remission | 1 months
  Proportion of patients in hematologic remission among all patients with morphological disease (NO CR) at enrollment

SECONDARY OUTCOMES:
Duration of MRD-negative remission | 2 years
  Duration of MRD-negative remission
Persistence/frequency of CD19 CAR T lymphocytes in peripheral (FC+qPCR) | 2 years
  Persistence/frequency of CD19 CAR T lymphocytes in peripheral (FC+qPCR)
Duration of B-cell aplasia | 5 years
  Duration of B-cell aplasia and hypogammaglobulinemia, time 0 - day of CD19-CAR T cells infusion
Overall survival | 5 years
  the probability of survival, time 0 - day of CD19-CAR T cells infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology and Immunology, Moscow, Russia

REFERENCES:
- [Derived] Maschan M, Caimi PF, Reese-Koc J, Sanchez GP, Sharma AA, Molostova O, Shelikhova L, Pershin D, Stepanov A, Muzalevskii Y, Suzart VG, Otegbeye F, Wald D, Xiong Y, Wu D, Knight A, Oparaocha I, Ferencz B, Roy A, Worden A, Kruger W, Kadan M, Schneider D, Orentas R, Sekaly RP, de Lima M, Dropulic B. Multiple site place-of-care manufactured anti-CD19 CAR-T cells induce high remission rates in B-cell malignancy patients. Nat Commun. 2021 Dec 10;12(1):7200. doi: 10.1038/s41467-021-27312-6. PMID 34893603